CLINICAL TRIAL: NCT06878118
Title: Prospective, Controlled, Randomised, Contralateral Wear, Dispensing Trial to Assess the Efficacy of Contact Lenses Using A.R.R.E.S.T.® Technology
Brief Title: The A.R.R.E.S.T.® Contact Lens Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: nthalmic Pty Ltd (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: nthal2024-03
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Myopia Progression
Keywords: axial length
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Intervention 1 (Active Comparator): Single vision contact lens
  Interventions: Device: Single-vision contact lens
- Assigned Intervention 2 (Experimental): A.R.R.E.S.T.® contact lens
  Interventions: Device: A.R.R.E.S.T.® contact lens

INTERVENTIONS:
Device: Single-vision contact lens — Standard single vision contact lens
  Arms: Assigned Intervention 1
Device: A.R.R.E.S.T.® contact lens — Contact lens with edge pattern
  Arms: Assigned Intervention 2

SUMMARY:
The goal of this clinical trial is to learn if contact lenses using Active Reconfiguration in Retinal Encoding of Spatio-Temporal (A.R.R.E.S.T.®) signal technology works to slow down the rate of myopia progression compared to single vision contact lenses in myopic children. The main questions it aims to answer are:

Do contact lenses using A.R.R.E.S.T.® technology slow down the rate of axial length growth? Do contact lenses using A.R.R.E.S.T.® technology slow down the rate of increase in myopic refractive error?

Researchers will compare contact lenses using A.R.R.E.S.T.® technology to a single vision contact lens.

Participants will:

Be randomly allocated to wear either contact lenses using A.R.R.E.S.T.® technology or single vision contact lenses.

Visit the clinic on seven occasions over a 12 month period.

DETAILED DESCRIPTION:
The aim of this clinical trial is to compare the rate of myopia progression as measured by change from dispensing, in axial length and the change from Baseline in the spherical equivalent cycloplegic autorefraction between a contact lens using A.R.R.E.S.T.® technology (test) and a single vision contact lens (control). Myopic children (7-15 years of age) will be randomly allocated to wear either test or control.

The overall trial duration, including follow-up period, is expected to be approximately 18 months. Each participant's duration is expected to be approximately 12 months.

The visits are Baseline, 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months.

All procedures performed at these visits are standard, non invasive clinical tests.

ELIGIBILITY:
Inclusion Criteria

* Be between 7 to 15 years old inclusive at time of enrolment.
* Have:

  * Read the Informed Assent.
  * Been explained the Informed Assent.
  * Indicated an understanding of the Informed Assent.
  * Signed the Informed Assent.
* Have their parent / legal guardian.

  * Read the Informed Consent.
  * Been explained the Informed Consent.
  * Indicated an understanding of the Informed Consent.
  * Signed the Informed Consent.
* Along with their parent/legal guardian, be capable of comprehending the nature of the study and be willing to adhere to the study requirements.
* Along with their parent/legal guardian, agree to maintain the visit and prescribed wearing schedule.
* Agree to wear the study contact lenses for a minimum of 5 days/week, 6 hours/day on days lenses are worn but not > 16 hours per day, and to remove lenses at night (i.e., daily wear only with no contact lens wear during sleep), for the duration of the study and to inform the investigator if their schedule is interrupted. Wearing time can be modified by the investigator for health reasons.
* Be in good general health, based on parent's/legal guardian's knowledge.
* Have best-corrected high contrast visual acuity of 0.10 logMAR (Snellen: 20/25, 6/7.6; Decimal: 0.80) or better in each eye.
* Meet the following criteria determined by cycloplegic autorefraction at Baseline:

  * -4.00 D ≤ spherical equivalent ≤ 0.75 D
  * -1.00 DC ≤ astigmatic component ≤ 0 DC
* Participants who fail astigmatism criterion with autorefraction pass astigmatism criterion if ≥ 0.75 D is measured with subjective refraction.

  * |Spherical equivalent anisometropia| ≤ 1.00 D.

Exclusion Criteria

* Participant in another study within 30 days prior to this study.
* Current or prior use of interventions intended for myopia control, including but not limited to:
* Optical devices:

  * Bifocal / multifocal spectacles.
  * Bifocal / multifocal contact lenses.
  * Orthokeratology.
* Pharmacological agents:

  * Atropine with a concentration > 0.01%.
  * Participants who have previously used 0.01% atropine are eligible for this study provided they agree not to use 0.01% atropine for at least 30 days before baseline and at any time during the study.
  * Pirenzepine.
* Participant born earlier than 30 weeks or weighed < 1500 g at birth.

  o A verbal report from the participant's parent / legal guardian is sufficient.
* Habitual use of a systemic or topical medication that may alter normal ocular findings / is known to affect a participant's ocular health / physiology either in an adverse or beneficial manner at enrolment and / or during the clinical trial.
* A known allergy to sodium fluorescein, benoxinate, proparacaine, tropicamide, or cyclopentolate.
* A known corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, ocular viral or fungal infections, or any other recurrent ocular infections.
* Strabismus as determined by cover test at distance (≥ 3 m) or near (40 cm) while wearing distance correction under non-cycloplegic conditions.
* Known ocular or systemic disease, such as but not limited to:

  * Diabetes.
  * Graves' disease.
  * Glaucoma.
  * Uveitis.
  * Scleritis.
  * Auto immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjogrens syndrome, and systemic lupus erythematosus.
  * Any ocular, systemic, or neuro-developmental conditions that could influence refractive development, such as but not limited to:
  * Persistent pupillary membrane.
  * Vitreous haemorrhage.
  * Cataract.
  * Central corneal scarring.
  * Eyelid haemangiomas.
  * Marfan's syndrome.
  * Down's syndrome.
  * Ehler's-Danlos syndrome.
  * Stickler's syndrome.
  * Ocular albinism.
  * Retinopathy of prematurity.
  * Keratoconus or irregular cornea.
* Biomicroscopic that contraindicate contact lens, such as but not limited to:

  * Neovascularisation or ghost vessels ≥ 1.5 mm in from limbus.
  * Any active anterior segment disease that contraindicates safe contact lens wear.
  * Clinically significant giant papillary conjunctivitis.
  * Clinically significant abnormalities of the anterior segment, lids, conjunctiva, sclera, or associated structures.
  * Allergic or seasonal conjunctivitis if the investigator believes it could significantly interfere with maintaining a specified wearing schedule.
* The investigator may, at their discretion, exclude anyone who they believe may not be able to fulfil the clinical trial requirements or it is believed to be in the participant's best interests.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-07-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Axial Length | Baseline, then1 month, 3 months, 6 months, 9 months, and 12 months after baseline
  Difference in change from baseline in axial length between each test and control.
Cycloplegic spherical equivalent autorefraction | Baseline, then 6 months, and 12 months after baseline
  Difference in change from Baseline in cycloplegic spherical equivalent autorefraction between each test and control.

SECONDARY OUTCOMES:
Visual performance as measured by high contrast visual acuity at 6 m | Baseline, then 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after baseline
  Difference in visual acuity between each test and control.
Visual performance as measured by a non validated questionnaire based on a 1-10 numeric rating scale | 1 month, 3 months, 6 months, 9 months, 12 months after baseline
  Difference in subjective visual performance between test and control after a minimum wear of one month.

CONTACTS AND LOCATIONS:
Locations (2):
- Wenzhou Medical University, Wenzhou, Zhejiang, China
- Optometry Clinic, Faculty of Health Science, Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.